CLINICAL TRIAL: NCT06183671
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multi-Part, Single and Multiple Ascending Dose Study of JX09 in Healthy Adult Participants
Brief Title: JX09 SAD/MAD in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ji Xing Pharmaceuticals Australia Pty Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Organization: Corxel Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JX09002
Record Dates: First submitted 2023-11-20; First posted 2023-12-27 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Resistant Hypertension
Keywords: Hypertension; Health Volunteer; Pharmacokinetic; Food effect
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Double-Blind, Placebo-Controlled, Multi-Part
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ascending Single Doses (Experimental): 48 participants, 6 single ascending dose (SAD) cohorts (Cohorts 1 to 6). Within each cohort, 8 participants will be randomized in a 6:2 ratio, 6 participants receiving JX09 and 2 receiving placebo
  Interventions: Drug: JX09 or placebo SAD
- Ascending Multiple Doses (Experimental): 32 participants, 4 multiple ascending dose (MAD) cohorts (Cohorts 7 to 10). Within each cohort, 8 participants will be randomized in a 6:2 ratio, 6 participants receiving JX09 and 2 receiving placebo
  Interventions: Drug: JX09 or placebo MAD
- Food Effect (Experimental): 12 participants,1 single-dose food effect (FE) cohort (Cohort 11), open-label, two-sequence, two-period, crossover design, participants will be randomly assigned to 1 of the 2 crossover sequences
  Interventions: Drug: JX09

INTERVENTIONS:
Drug: JX09 or placebo SAD — For Part 1 SAD: JX09/placebo in capsule will be administered as a single oral dose. The nominal dose escalation scheme for the cohorts is 1, 3, 10, 30, 100, and 300 mg.
  Arms: Ascending Single Doses
Drug: JX09 or placebo MAD — For Part 2 MAD: JX09/placebo in capsule will be administered for 11 days (once daily) The nominal dose escalation scheme for the cohorts is 2, 5, 10 and 20 mg.
  Arms: Ascending Multiple Doses
Drug: JX09 — For Part 3 FE: JX09 in capsule will be administered as a two single oral doses separated by 15 days. The nominal dose is 10 mg.
  Arms: Food Effect

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, multi-part, single and multiple ascending dose study in healthy adult to test the safety, tolerability, pharmacokinetics, pharmacodynamics, and food effect of JX09 when administered to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 55 years (inclusive)
* In good health as deemed by the Investigator through a medical evaluation, including medical history, physical examination, and laboratory tests
* Body mass index (BMI) between 18 and 32 kg/m2, with a minimum weight of 50 kg at Screening

Exclusion Criteria:

* Clinically significant oncologic, infectious, cardiovascular, pulmonary, hepatic, gastrointestinal, hematologic, metabolic, endocrine, neurologic, immunologic, renal, psychiatric, or other condition that in the opinion of the Investigator or Medical Monitor would make is unsafe for the participant to join the study or fulfill its requirements.
* A clinical abnormality or abnormal laboratory parameter(s) in the opinion of the Investigator or Medical Monitor is likely to introduce additional risk or will affect data interpretation.
* Postural tachycardia or hypotension.
* Female of childbearing potential who is pregnant, lactating, or planning to become pregnant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events and serious adverse events in health subjects. | For SAD cohort,11 days, from Day 1 to Day 11; for MAD cohort,21 days, from Day 1 to Day 21; for food effect cohort,26 days, from Day 1 to Day 26
  The number of AEs and SAEs by using Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Clinically significant change from baseline in physical examinations in health subjects | For SAD cohort,11 days, from Day 1 to Day 11; for MAD cohort,21 days, from Day 1 to Day 21; for food effect cohort,26 days, from Day 1 to Day 26
  The number of events that clinically significant change from baseline in physical examinations by measuring general appearance, head, ears, eyes, nose, throat, dentition, thyroid, chest, abdomen, skin, neurological extremities, etc.
Clinically significant change from baseline in vital signs in health subjects | For SAD cohort,11 days, from Day 1 to Day 11; for MAD cohort,21 days, from Day 1 to Day 21; for food effect cohort,26 days, from Day 1 to Day 26
  The number of events that clinically significant change from baseline in vital signs by measuring heart rate, blood pressure, temperature, and respiratory rate.
Clinically significant change from baseline in electrocardiograms in health subjects | For SAD cohort,11 days, from Day 1 to Day 11; for MAD cohort,21 days, from Day 1 to Day 21; for food effect cohort,26 days, from Day 1 to Day 26
  The number of events that clinically significant change from baseline in electrocardiograms by measuring heart rate, PR, QRS, QT and QTc interval.
Clinically significant change from baseline in clinical laboratory tests in health subjects | For SAD cohort,11 days, from Day 1 to Day 11; for MAD cohort,21 days, from Day 1 to Day 21; for food effect cohort,26 days, from Day 1 to Day 26
  The number of events that clinically significant change from baseline in clinical laboratory tests by measuring clinical chemistry panel, complete blood count and coagulation.

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters after a single ascending dose in health subjects | From Day 1 to Day 11
  Area under the Concentration time Curve from Time 0 to the Last Measurable Concentration (AUC0-t) by measuring blood plasma
Plasma pharmacokinetic parameters after a single ascending dose in health subjects | From Day 1 to Day 11
  Area under the Concentration-time Curve from Time 0 to 24 hour (AUC0-24) by measuring blood plasma
Plasma pharmacokinetic parameters after a single ascending dose in health subjects | From Day 1 to Day 11
  Area under the Concentration-time Curve from Time 0 to Infinity (AUC0-inf) by measuring blood plasma
Plasma pharmacokinetic parameters after a single ascending dose in health subjects | From Day 1 to Day 11
  Peak plasma concentration (CMAX) by measuring blood plasma
Plasma pharmacokinetic parameters after a single ascending dose in health subjects | From Day 1 to Day 11
  Time of maximum concentration (TMAX) by measuring blood plasma
Plasma pharmacokinetic parameters after multiple ascending dose in health subjects | On day 1 and day 11
  Peak plasma concentration (CMAX) by measuring blood plasma
Plasma pharmacokinetic parameters after multiple ascending dose in health subjects | On day 1 and day 11
  Time of maximum concentration (TMAX) by measuring blood plasma
Plasma pharmacokinetic parameters after multiple ascending dose in health subjects | On day 1 and day 11
  Area under the Concentration time Curve from Time 0 to the Last Measurable Concentration (AUC0-t) by measuring blood plasma
Plasma pharmacokinetic parameters after multiple ascending dose in health subjects | On day 1 and day 11
  Area under the Concentration-time Curve from Time 0 to 24 hour (AUC0-24) by measuring blood plasma
Plasma pharmacokinetic parameters after multiple ascending dose in health subjects | From day 2 to day 11
  Concentration at end of dosing interval by measuring blood plasma
Plasma pharmacokinetic parameters in health subjects under fed and fasted conditions | From day 1 to day 5 and on day 11, From day 16 to day 20 and day 26
  Area under the Concentration time Curve from Time 0 to the Last Measurable Concentration (AUC0-t) by measuring blood plasma
Plasma pharmacokinetic parameters in health subjects under fed and fasted conditions | From day 1 to day 5 and on day 11, From day 16 to day 20 and day 26
  Area under the Concentration-time Curve from Time 0 to 24 hour (AUC0-24) by measuring blood plasma
Plasma pharmacokinetic parameters in health subjects under fed and fasted conditions | From day 1 to day 5 and on day 11, From day 16 to day 20 and day 26
  Area under the Concentration-time Curve from Time 0 to Infinity (AUC0-inf) by measuring blood plasma
Urine pharmacokinetic parameters after multiple ascending dose in health subjects | on day 1 and day 11
  Cumulative amount of drug excreted by measuring urine
Urine pharmacokinetic parameters after multiple ascending dose in health subjects | on day 1 and day 11
  Fraction of the dose excreted renally by measuring urine
Urine pharmacokinetic parameters after multiple ascending dose in health subjects | on day 1 and day 11
  Renal clearance by measuring urine
Plasma pharmacodynamic parameters after a single ascending dose or multiple ascending dose in health subjects | From Day -1 to Day 5 and Day 11 for SAD cohort and from Day -2 to Day 1 and from Day 7 to Day 15 and Day 21 for MAD cohort
  Change from baseline of aldosterone by measuring blood plasma
Plasma pharmacodynamic parameters after a single ascending dose or multiple ascending dose in health subjects | From Day -1 to Day 5 and Day 11 for SAD cohort and from Day -2 to Day 1 and from Day 7 to Day 15 and Day 21 for MAD cohort
  Change from baseline of cortisol by measuring blood plasma
Plasma pharmacodynamic parameters after a single ascending dose or multiple ascending dose in health subjects | From Day -1 to Day 5 and Day 11 for SAD cohort and from Day -2 to Day 1 and from Day 7 to Day 15 and Day 21 for MAD cohort
  Change from baseline of corticosterone by measuring blood plasma
Urine pharmacodynamic parameters after a single ascending dose or multiple ascending dose in health subjects | On Day 1 for SAD cohort and on Day -1 and 11 for MAD cohort
  Change from baseline of sodium by measuring 24-hour urine level
Urine pharmacodynamic parameters after a single ascending dose or multiple ascending dose in health subjects | On Day 1 for SAD cohort and on Day -1 and 11 for MAD cohort
  Change from baseline of potassium by measuring 24-hour urine level
Urine pharmacodynamic parameters after a single ascending dose or multiple ascending dose in health subjects | On Day 1 for SAD cohort and on Day -1 and 11 for MAD cohort
  Change from baseline of aldosterone by measuring 24-hour urine level
Urine pharmacodynamic parameters after a single ascending dose or multiple ascending dose in health subjects | On Day 1 for SAD cohort and on Day -1 and 11 for MAD cohort
  Change from baseline of cortisol by measuring 24-hour urine level

CONTACTS AND LOCATIONS:
Overall Officials: Sam Francis, MD, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Australia